CLINICAL TRIAL: NCT01093651
Title: A Blinded Randomized Controlled Pilot Immunologic and Virologic Safety Trial of an FDA-approved DPPIV-inhibitor in HIV+ Men and Women
Brief Title: Dipeptidyl Peptidase-4 Inhibition and Immune Function in HIV
Acronym: DPPIVinHIV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Campbell Foundation (Other)
Responsible Party: Principal Investigator, Kevin Yarasheski, PhD, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KEY03222010
Record Dates: First submitted 2010-03-23; First posted 2010-03-26 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DPPIV inhibition (Experimental): Four to six months of sitagliptin administration (100mg/d) to people living with HIV-1 who have well-controlled immunologic (CD4+ T-cell count >350 cells/µL) and virologic (plasma HIV RNA <50 copies/mL) status.
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Four to six months of placebo to people living with HIV-1 who have well-controlled immunologic (CD4+ T-cell count >350 cells/µL) and virologic (plasma HIV RNA <50 copies/mL) status.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg sitagliptin daily for 4-6 months
  Arms: DPPIV inhibition
Drug: Placebo — Daily placebo for 4-6 months
  Arms: Placebo

SUMMARY:
We will test the safety of a new class of anti-diabetes compounds (DPPIV-inhibitors) in people living with HIV. Future trials will examine efficacy for treating diabetes and reducing cardiovascular disease risk in people living with HIV.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV)-infection and treatment with antiretroviral therapies are associated with several cardiometabolic risk factors; insulin resistance, diabetes, dyslipidemia, central adiposity, that increase risk for MI and stroke. A new class of drugs used to treat type 2 diabetes has been introduced; Dipeptidyl peptidase-IV (DPPIV)-inhibitors (Januvia®, Onglyza®, alogliptin). Dipeptidyl peptidase-IV (DPPIV)-inhibition could be a safe and effective therapy for HIV-associated insulin resistance and diabetes. However, no safety data exist. The research question is: If HIV+ adults with stable immunologic (CD4+ T-cell count >350 cells/μL) and virologic (plasma HIV RNA <50 copies/mL) function are given a DPPIV-inhibitor would their CD4+ T-cell count and plasma HIV RNA level increase, decrease, or stay the same? Theoretically, DPPIV-inhibition could enhance their immune system by increasing SDF-1α levels; a potent inhibitor of HIV-entry into T-cells, or harm the HIV+ immune system by inactivating CD26 on immune cells. We hypothesize that DPPIV-inhibition will not harm the immune system in HIV+ people. We propose a blinded randomized controlled pilot safety trial of an FDA-approved DPPIV-inhibitor in virologically- and immunologically-stable HIV+ men and women. We will monitor CD4+ T-cell count, plasma HIV RNA levels, immune activation markers, and safety outcomes (lipid/lipoprotein profiles, blood pressure, kidney and liver function) during 4-6 months of DPPIV-inhibitor exposure vs placebo in 20 HIV+ adults. If safety is confirmed, the efficacy of DPPIV-inhibition in HIV+ with insulin resistance will be tested in future trials that examine potential glucoregulatory and cardiovascular benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Thirty 18-65 yr old HIV-infected men and women (with source documentation of HIV status) who are stable on any antiretroviral therapy (cART) regimen
2. Have stable (at least the past 12-months) immunologic (>350 CD4+ T-cells/µL) and virologic (<50 copies HIV RNA/mL) status.
3. BMI 18-42kg/m2;
4. Normal blood chemistry for at least 1 month prior to enrollment;
5. Platelet count > 30,000/mm3, absolute neutrophil count >750/mm3, transaminases < 2.5x the upper limit of normal (ULN).
6. Long-term non-progressors (not on ART) are not eligible.

Exclusion Criteria:

1. CD4+ T-cell count <350 cells/µL or detectable plasma HIV RNA (>50 copies HIV RNA/mL) within the past 12-months. During the study, if CD4+ T-cell count declines by >100 cells/µL, or if plasma HIV RNA becomes detectable (>50 copies HIV RNA/mL after repeat analysis 2wks apart), and the participant denies any lapse in their anti-HIV medication regimen, the study medication will be stopped and an adverse event documented. If at any time during the study, two participants experience a reduction in T-cell count >100 cells/µL, or their plasma HIV RNA levels become detectable (>50 copies HIV RNA/mL after repeat analysis 2wks apart), and they are confirmed (by unblinding) to have received sitagliptin, the study will be stopped for serious safety concerns.
2. Systemic, secondary or opportunistic infection within past 12-months.
3. Fasting glucose intolerance (FBG >100mg/dL), fasting hyperinsulinemia (>15µU/mL), or fasting insulin resistance (Homeostasis model for insulin resistance (HOMA) >3.0). Any agents that might alter glucose metabolism (insulin, TZDs, metformin, glucocorticoids, sulfonylurea, corticosteroids, megace, rhGH, GH-secretagogue) during the 3 months prior to enrollment or at any time during enrollment. Volunteers with T2DM, IDDM or diabetic ketoacidosis will not be enrolled.
4. History of serious CV disease or NYHA Functional Class III or IV, (e.g., recent MI, unstable angina, edema, CHF, CAD, CABG, valve disease (murmur), stroke, uncontrolled high blood pressure (resting >160/95 mmHg), irregular heart rhythm, resting ST-segment depression >1mm). Treatment with medications for a CV condition (cardiac glycosides α- or ß-blockers). Some antihypertensive medications (calcium-channel blocker, diuretic, angiotensin II receptor blockers (ARB), angiotensin converting enzyme inhibitors (ACE)) will be permitted.
5. Moderate to severe renal insufficiency. Serum creatinine >1.7 mg/dL (men) >1.5 mg/dL (women).
6. Known allergy or hypersensitivity to DPPIV-inhibitors.
7. Plan to change anti-HIV medication regimen or prophylaxis for opportunistic infection within 6-months of starting study.Transitions among efavirenz-based regimens will be allowed (e.g., Efavirenz + lamivudine + zidovudine (combivir) to Efavirenz + emtricitabine + tenofovir (Atripla)).
8. Lipid-lowering medications are permitted (fibrate or statin or niacin), but must be stable on that agent for at least 3 months prior to enrollment. Lipid-lowering agents cannot be started during the treatment period.
9. Chronic hepatitis B infection (HB surface antigen positive). Active hepatitis C infection (detectable Hep C RNA). Those who have cleared hepatitis B or C infection are eligible.
10. Hematocrit <34% in men or <25% in women with symptoms (fatigue, "tired-legs", shortness of breath). Hemoglobin <10 gm/100ml with symptoms.
11. Nausea, vomiting, diarrhea (>4 loose stools/day) that are unresponsive to treatment. History of eating disorder or significant GI-disease.
12. Pregnant or nursing mothers. Women must agree to use an acceptable form of birth control during the study. If birth control pills are used, the woman must be stable on these medications for at least 6 months prior to enrollment.
13. Active malignancy or treatment with chemotherapeutic agents or radiation therapy (within past 12 months).
14. >10% unintentional body weight loss during the 12 months prior to enrollment.
15. "Blinded" investigational drugs/medications during the 3 months prior to enrollment that will not be unblinded before enrollment. Open-label investigational drugs are permitted (within past 3 months, no plan to stop during enrollment and not known to affect glucose, lipid, adipose tissue or liver metabolism).
16. Over the counter agents that might alter glucose, lipid, or adipose tissue metabolism (e.g., creatine monohydrate, chromium picolinate, amino acid/protein supplements, medium- or long-chain fatty acids) within 1 month of enrollment. These supplements are not permitted during the treatment period.
17. Reduced cognitive function/unable to provide voluntary informed consent. Prisoners are excluded.
18. Active substance abuse that the physician-scientist believes may compromise safety, compliance, or interfere with study drug or data interpretation.
19. Any cytokine or anti-cytokine therapy during 3 months prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Yarasheski, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Goodwin SR, Reeds DN, Royal M, Struthers H, Laciny E, Yarasheski KE. Dipeptidyl peptidase IV inhibition does not adversely affect immune or virological status in HIV infected men and women: a pilot safety study. J Clin Endocrinol Metab. 2013 Feb;98(2):743-51. doi: 10.1210/jc.2012-3532. Epub 2012 Dec 21. PMID 23264399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-infected adults (18 - 65 years old) were recruited from the AIDS Clinical Trials Unit and the Infectious Diseases Clinic at Washington University School of Medicine. Thirty-one candidates were screened and 20 were enrolled; all participants were HIV positive but were otherwise healthy with stable immunologic and virologic status on HAART.
Pre-assignment Details: Twenty participants were randomized to n=10 placebo or n=10 sitagliptin (Januvia(R)). Eleven volunteers were screened and found ineligible (see eligibility criteria), or did not choose to participate in the study.
Groups:
- Placebo: Four months of placebo to people living with HIV-1 who have well-controlled immunologic (CD4+ T-cell count >350 cells/µL) and virologic (plasma HIV RNA <50 copies/mL) status.
  Placebo : Daily placebo for 4 months
- DPPIV Inhibition: Four months of sitagliptin administration (100mg/d) to people living with HIV-1 who have well-controlled immunologic (CD4+ T-cell count >350 cells/µL) and virologic (plasma HIV RNA <50 copies/mL) status.
  Sitagliptin : 100 mg sitagliptin daily for 4 months
Period: Overall Study
Arm/Group | Placebo | DPPIV Inhibition
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DPPIV Inhibition | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (15) | 36 (9) | 38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: CD4+ T-cell Count
Time Frame: Monthly for 4 months
Population: CD4+ T-cell count
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Placebo | DPPIV Inhibition
Number analyzed (Participants) | 10 | 10
cells/µL
  Baseline | 602 (91) | 648 (185)
  Week 4 | 689 (153) | 750 (225)
  Week 8 | 696 (194) | 656 (207)
  Week 12 | 686 (167) | 706 (168)
  Week 16 | 681 (151) | 636 (173)
Statistical Analysis 1: Comparison: Placebo vs DPPIV Inhibition; The main effect analysis was applied to both rows (timepoint) and categories (groups). It used linear mixed models to simultaneously assess differences in CD4+ T-cell count between the DPP4 inhibitor and placebo groups (categories) over time (rows). Pairwise post-hoc contrasts were performed to assess the between and within group differences in outcome measures at each time point; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05. The main effect analysis for CD4+ T-cell count over time and between the 2 groups did not achieve p<0.05 (not statistically significant); Study subject was included in these models as a random variable to account for within-participant correlation

2. Primary Outcome: Plasma HIV Viremia (Viral Load)
Description: Percentage of participants with plasma HIV RNA copy number less than 48 copies/mL
Time Frame: Monthly for 6 months
Measure: Number; unit: percentage of participants below 48 c/mL
Arm/Group | Placebo | DPPIV Inhibition
Number analyzed (Participants) | 10 | 10
percentage of participants below 48 c/mL
  Baseline | 100 | 100
  Week 4 | 100 | 100
  Week 8 | 100 | 100
  Week 12 | 100 | 100
  Week 16 | 100 | 100
  Week 24 | 100 | 100
Statistical Analysis 1: Comparison: Placebo vs DPPIV Inhibition; The main effect analysis was applied to both rows (timepoint) and categories (groups). It used linear mixed models to simultaneously assess differences in plasma HIV RNA copy number/mL between the DPP4 inhibitor and placebo groups (categories) over time (rows). Pairwise post-hoc contrasts were performed to assess the between and within group differences in outcome measures at each time point; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05. The main effect analysis for plasma HIV RNA copy number/mL over time and between the 2 groups did not achieve p<0.05 (not statistically significant)

3. Secondary Outcome: Soluble TNFR2; Serum Biomarkers of Immune Activation
Description: serum soluble tumor necrosis factor receptor-2 concentration
Time Frame: Baseline, week 8, week 16
Population: sTNFR2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | DPPIV Inhibition
Number analyzed (Participants) | 10 | 10
pg/mL
  Baseline | 2220 (389) | 2436 (431)
  week 8 | 2218 (411) | 2617 (638)
  week 16 | 2279 (415) | 2388 (449)
Statistical Analysis 1: Comparison: Placebo vs DPPIV Inhibition; The main effect analysis was applied to both rows (timepoint) and categories (groups). It used linear mixed models to simultaneously assess differences in serum TNFR2 levels between the DPP4 inhibitor and placebo groups (categories) over time (rows). Pairwise post-hoc contrasts were performed to assess the between and within group differences in outcome measures at each time point; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05. The main effect analysis for serum TNFR2 levels over time and between the 2 groups did not achieve p<0.05 (not statistically significant)

4. Secondary Outcome: SDF1α; Serum Biomarkers of Immune Activation
Description: serum stromal cell-derived factor-1α concentration
Time Frame: Baseline, week 8, week 16
Population: SDF1α
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | DPPIV Inhibition
Number analyzed (Participants) | 10 | 10
pg/mL
  Baseline | 2327 (304) | 2378 (441)
  week 8 | 2313 (364) | 1208 (605)
  week 16 | 2309 (400) | 1277 (490)
Statistical Analysis 1: Comparison: Placebo vs DPPIV Inhibition; The main effect analysis was applied to both rows (timepoint) and categories (groups). It used linear mixed models to simultaneously assess differences in serum SDF1α levels between the DPP4 inhibitor and placebo groups (categories) over time (rows). Pairwise post-hoc contrasts were performed to assess the between and within group differences in outcome measures at each time point; Test type: Superiority or Other; p < 0.0002, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05. The main effect analysis for SDF1-alpha levels over time and between the 2 groups achieved p<0.0002

5. Secondary Outcome: RANTES; Serum Biomarkers of Immune Activation
Description: serum Regulated on Activation, Normal T cell Expressed and Secreted concentration
Time Frame: Baseline, week 8, week 16
Population: RANTES
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | DPPIV Inhibition
Number analyzed (Participants) | 10 | 10
ng/mL
  Baseline | 80.8 (23.2) | 64.4 (37.2)
  week 8 | 85.3 (27.7) | 68.5 (43.0)
  week 16 | 74.9 (27.8) | 62.8 (32.3)
Statistical Analysis 1: Comparison: Placebo vs DPPIV Inhibition; The main effect analysis was applied to both rows (timepoint) and categories (groups). It used linear mixed models to simultaneously assess differences in serum RANTES levels between the DPP4 inhibitor and placebo groups (categories) over time (rows). Pairwise post-hoc contrasts were performed to assess the between and within group differences in outcome measures at each time point; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05. The main effect analysis for serum RANTES levels over time and between the 2 groups did not achieve p<0.05 (not statistically significant)

6. Secondary Outcome: Oral Glucose Tolerance
Description: Area under the 75-gr oral glucose tolerance curve (AUCg) based on plasma glucose values measured at 0, 30, 60, 90, and 120 mins post-glucose challenge.
Time Frame: Baseline, week 8, week 16
Measure: Mean (Standard Deviation); unit: mg*min/mL
Arm/Group | Placebo | DPPIV Inhibition
Number analyzed (Participants) | 10 | 10
mg*min/mL
  Baseline AUCg | 142.5 (26.6) | 145.6 (32.5)
  Week 8 AUCg | 158.0 (26.7) | 133.6 (24.6)
  Week 16 AUCg | 157.5 (23.2) | 142.5 (21.5)
Statistical Analysis 1: Comparison: Placebo vs DPPIV Inhibition; The main effect analysis was applied to both rows (timepoint) and categories (groups). It used linear mixed models to simultaneously assess differences in area under the glucose tolerance curves between the DPP4 inhibitor and placebo groups (categories) over time (rows). Pairwise post-hoc contrasts were performed to assess the between and within group differences in outcome measures at each time point; Test type: Superiority or Other; p < 0.04, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05. The main effect analysis for area under the glucose tolerance curve over time and between the 2 groups achieved p<0.04

7. Secondary Outcome: Self-reported Symptoms
Description: Cumulative number of self-reported symptoms based on the Division of AIDS Grading Scale for the Severity of Adult Adverse Events (0-4 scale where 0 is no new symptoms, 4 is serious adverse event or toxicity)
Time Frame: Monthly for 4 months
Population: Cumulative frequency over 16 weeks of any self-reported symptoms on the DAIDS scale
Measure: Number; unit: total number of self reported symptoms
Arm/Group | Placebo | DPPIV Inhibition
Number analyzed (Participants) | 10 | 10
total number of self reported symptoms
  Hypoglycemia symptoms | 1 | 3
  GI symptoms | 8 | 3
  Upper respiratory symptoms | 10 | 5
  Generalized fatigue | 5 | 2
  Headache | 5 | 4
  Other (e.g., rash, muscle pain, mood change) | 6 | 5
Statistical Analysis 1: Comparison: Placebo vs DPPIV Inhibition; Kruskal-Wallis non-parametric test of cell frequencies; Test type: Superiority or Other; p > 0.05, Kruskal-Wallis — The a priori threshold for statistical significance was p<0.05. The non-paramteric test for adverse event cummulative frequency between the 2 groups did not achieve p<0.05 (not statistically significant)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: SAE or AE Any self reported symptom that was graded greater than 2 on the DAIDS severity scale during the 16 week period. These were reported as a serious or adverse event or toxicity.
  Other adverse event: Any self-reported symptom that was graded less than or equal to 2 (DAIDS scale) during the 16 week period;these are not serious adverse events.
Arm/Group | Placebo | DPPIV Inhibition
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | DPPIV Inhibition (N=10)
Hypoglycemia symptoms (Metabolism and nutrition disorders) | 1 (1) | 2 (3) — Not SAE; severity graded less than 2 on DAIDS
Gastrointestinal symptoms (Gastrointestinal disorders) | 5 (8) | 2 (3) — Not SAE; severity graded less than 2 on DAIDS
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 3 (5) — Not SAE; severity graded less than 2 on DAIDS
Generalized fatigue (General disorders) | 3 (5) | 1 (2) — Not SAE; severity graded less than 2 on DAIDS
Headache (General disorders) | 4 (5) | 2 (4) — Not SAE; severity graded less than 2 on DAIDS
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) — Not SAE; severity graded less than 2 on DAIDS
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Not SAE; severity graded less than 2 on DAIDS
Mood change (Psychiatric disorders) | 2 (3) | 2 (3) — Not SAE; severity graded less than 2 on DAIDS

LIMITATIONS AND CAVEATS:
Potential for type 2 error given small sample size. But, study was powered to detect significant decline in CD4 count. Measures of monocyte and lymphocyte activation should be conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No